CLINICAL TRIAL: NCT00389857
Title: Annual Study for Serum Collection and Evaluation of Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Influenza Virus Vaccine (2006-2007 Formulation)
Brief Title: Trial to Collect Safety Data and Sera for Immunogenicity Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC34
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Results first posted 2009-03-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Influenza Virus Vaccine; Fluzone®
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine-naive group (Experimental): Participants have never received Influenza virus vaccine in the past. They will receive a single dose of Fluzone vaccine on Day 0 and Day 28, respectively.
  Interventions: Biological: Influenza Virus Vaccine (Fluzone®)
- Influenza vaccine-primed group (Experimental): Participants have received Influenza virus vaccine in the past. They will receive a single dose of Fluzone vaccine on Day 0.
  Interventions: Biological: Influenza Virus Vaccine (Fluzone®)

INTERVENTIONS:
Biological: Influenza Virus Vaccine (Fluzone®) — 0.25 mL, Intramuscular (infant/children dose)
  Other Names: Fluzone®
  Arms: Influenza vaccine-naive group
Biological: Influenza Virus Vaccine (Fluzone®) — 0.25 mL, Intramuscular (infant/children dose)
  Other Names: Fluzone®
  Arms: Influenza vaccine-primed group

SUMMARY:
To provide Centers for Biologics Evaluation and Research (CBER) with sera collected from healthy children receiving the 2006-2007 formulation of the inactivated, split-virion influenza vaccine Fluzone® for further study by the Food and Drug Administration (FDA), Center for Disease Control and Prevention (CDC) and World Health Organization (WHO).

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged ≥ 6 months (24 weeks) to < 36 months (3rd birthday).
* Participant is considered to be in good health on the basis of reported medical history and limited physical examination.
* Participant is available for the duration of the study.
* Parent/legal acceptable representative is willing and able to provide informed consent.
* Parent/legal acceptable representative is willing and able to meet protocol requirements.
* Born at full term of pregnancy (≥ 37 weeks) with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* Reported allergy to egg proteins, chicken proteins, or any other constituent of the vaccine.
* An acute illness with or without fever (For infants/toddlers: temperature

  ≥ 100.4 °F rectal; For children: temperature ≥ 99.5 °F oral/axillary) in the 72 hours preceding enrollment in the trial (Enrollment may be deferred).
* Clinically significant findings in vital signs or review of systems (investigator judgment; defer or exclude).
* Participation in any other interventional clinical trial within 30 days prior to enrollment up to termination of the subject's participation in the study.
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Personal or immediate family history of congenital immune deficiency.
* Developmental delay, neurologic disorder, or seizure disorder.
* Chronic medical, congenital, or developmental disorder.
* Known human immunodeficiency virus (HIV)-positive mother.
* Prior personal history of Guillain-Barré syndrome.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 13 October to 13 December 2006, at a single site in the US.
Pre-assignment Details: A total of 31 subjects that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Influenza Vaccine-Naive Group: Participants have never received Influenza virus vaccine in the past. They received a single dose of Fluzone® vaccine on Day 0 and Day 28, respectively.
- Influenza Vaccine-Primed Group: Participants have received Influenza virus vaccine in the past. They received a single dose of Fluzone® vaccine on Day 0.
Period: Overall Study
Arm/Group | Influenza Vaccine-Naive Group | Influenza Vaccine-Primed Group
Started | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine-Naive Group | Influenza Vaccine-Primed Group | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 17 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 15.4 (7.40) | 29.3 (6.55) | 23.0 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibodies Before and After Fluzone® Vaccination
Description: GMTs and their 95% Confidence Interval are presented for each of the 3 antigens in the Fluzone vaccine 2006-2007 Pediatric formulation.
  Post-dose 1 (Influenza vaccine-primed group); Post-dose 2 (Influenza vaccine-naive group)
Time Frame: 14 days post-vaccination
Population: Geometric mean titers were evaluated in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Influenza Vaccine-Naive Group: Subjects have never received Influenza virus vaccine
- Influenza Vaccine-Primed Group: Subjects have received Influenza virus vaccine in the past
Arm/Group | Influenza Vaccine-Naive Group | Influenza Vaccine-Primed Group
Number analyzed (Participants) | 13 | 12
Titer
  H1N1 Flu A/New Caledonia/20/99 - Pre | 5.36 [4.83 to 5.95] | 15.1 [6.51 to 34.8]
  H1N1 Flu A/New Caledonia/20/99 - Post | 169 [77.5 to 367] | 135 [61.9 to 293]
  H3N2 Flu A/Wisconsin/67/2005 - Pre | 13.7 [2.97 to 62.8] | 22.0 [8.27 to 58.4]
  H3N2 Flu A/Wisconsin/67/2005 - Post | 806 [316 to 2056] | 698 [400 to 1218]
  Flu B/Malaysia Split/2506/2004 - Pre | 5.55 [4.92 to 6.25] | 6.23 [4.71 to 8.25]
  Flu B/Malaysia Split/2506/2004 - Post | 234 [107 to 511] | 54.8 [20.9 to 144]

2. Other Pre Specified Outcome: Number of Participants Who Had Solicited Injection Site and Systemic Reactions Post-vaccination 1.
Description: Solicited injection site reactions: Erythema, swelling, tenderness for infants/toddlers, and pain for children Solicited systemic reactions: For infants/toddler: fever (temperature), irritability, abnormal crying, drowsiness, lost appetite, vomiting; For children: fever (temperature), headache, malaise, myalgia).
Time Frame: 0 to 3 days post-vaccination 1
Population: Safety analysis was on all enrolled and vaccinated participants, intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Influenza Vaccine-Naive Group | Influenza Vaccine-Primed Group
Number analyzed (Participants) | 14 | 17
Participants
  Any Solicited Injection Site Reaction Post-dose 1 | 3 | 6
  Any injection site Tenderness | 3 | 2
  Grade 3 injection site Tenderness-reduced movement | 0 | 0
  Any injection site Pain | 0 | 4
  Grade 3 injection site Pain (Incapacitating) | 0 | 0
  Any injection site Redness | 2 | 1
  Grade 3 injection site Redness (≥ 5.0 cm) | 0 | 0
  Any injection site Swelling | 1 | 0
  Grade 3 injection site Swelling (≥ 5.0 cm) | 0 | 0
  Any Solicited Systemic Reaction Post-dose 1 | 7 | 7
  Any Fever | 0 | 1
  Grade 3 Fever (>103.1°F) | 0 | 0
  Any Vomiting (Per 24 hours) | 2 | 0
  Grade 3 Vomiting (≥ 6 episodes) | 0 | 0
  Any Abnormal Crying | 3 | 2
  Grade 3 Abnormal Crying (> 3 hours) | 0 | 0
  Any Drowsiness | 1 | 1
  Grade 3 Drowsiness (Sleeping most time) | 0 | 0
  Any Loss of Appetite | 1 | 2
  Grade 3 Loss of Appetite (Refuses ≥ 3 feeds) | 0 | 0
  Any Irritability | 5 | 2
  Grade 3 Irritability (Inconsolable) | 0 | 0
  Any Headache | 0 | 3
  Grade 3 Headache (Prevented daily activities) | 0 | 0
  Any Myalgia | 1 | 1
  Grade 3 Myalgia (Prevented daily activities) | 0 | 0
  Any Malaise | 2 | 3
  Grade 3 Malaise (Prevented daily activities) | 0 | 0

3. Other Pre Specified Outcome: Number of Participants Who Had Solicited Injection Site and Systemic Reactions Post-vaccination 2.
Description: Solicited injection site reactions: Erythema, swelling, tenderness for infants/toddlers, and pain for children Solicited systemic reactions: For infants/toddler: fever (temperature), irritability, abnormal crying, drowsiness, lost appetite, vomiting; For children: fever (temperature), headache, malaise, myalgia).
  Note: Influenza vaccine-primed group did not receive vaccination 2
Time Frame: 0 to 3 days post-vaccination 2
Population: Safety analysis was on all enrolled and vaccinated participants, intend to treat population.
  Influenza vaccine-primed group did not received vaccination 2
Measure: Number; unit: Participants
Arm/Group | Influenza Vaccine-Naive Group | Influenza Vaccine-Primed Group
Number analyzed (Participants) | 14 | 0
Participants
  Any solicited injection site reaction Post-dose 2 | 4 |
  Any injection site Tenderness | 4 |
  Grade 3 injection site Tenderness-reduced movement | 0 |
  Any injection site Pain | 0 |
  Grade 3 injection site Pain (incapacitating) | 0 |
  Any injection site Redness | 3 |
  Grade 3 injection site Redness (≥ 5.0 cm) | 0 |
  Any injection site Swelling | 1 |
  Grade 3 injection site Swelling (≥ 5.0 cm) | 0 |
  Any solicited systemic reaction Post-dose 2 | 6 |
  Any Fever | 1 |
  Grade 3 Fever (> 103.1ºF) | 0 |
  Any Vomiting (per 24 hours) | 2 |
  Grade 3 Vomiting (≥ 6 episodes) | 0 |
  Any abnormal Crying | 4 |
  Grade 3 abnormal Crying (> 3 hours) | 0 |
  Any Drowsiness | 3 |
  Grade 3 Drowsiness (sleeping most time) | 0 |
  Any Loss of appetite | 5 |
  Grade 3 Loss of appetitie (refuses 3 feeds) | 0 |
  Any Irritability | 5 |
  Grade 3 Irritability (inconsolable) | 0 |
  Any Headache | 0 |
  Grade 3 Headache (prevents daily activities) | 0 |
  Any Myalgia | 0 |
  Grade 3 Myalgia (prevents daily activities) | 0 |
  Any Malaise | 0 |
  Grade 3 Malaise (prevents daily activities) | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 14 days post-vaccination (Influenza vaccine-primed) and for 42 days post-vaccination (Influenza vaccine-naive) participants.
Arm/Group | Influenza Vaccine-Naive Group | Influenza Vaccine-Primed Group
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 9/14 | 7/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine-Naive Group (N=14) | Influenza Vaccine-Primed Group (N=17)
Injection site tenderness (General disorders) | 4 | 2
Injection site pain (General disorders) | 0 | 4
Injection site redness (General disorders) | 3 | 1
Injection site swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Vomiting NOS (Gastrointestinal disorders) | 2 | 0
Crying (Psychiatric disorders) | 4 | 2
Somnolence (Nervous system disorders) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 2
Irritability (Psychiatric disorders) | 6 | 2
Headache (Nervous system disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Malaise (General disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Teething (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Irritability (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications